CLINICAL TRIAL: NCT01707940
Title: Relative Bioavailability of a Single Oral Dose of BI 144807 (Oral Solution) When Administered Alone or in Combination With Multiple Oral Doses of Ketoconazole (200 mg Tablet) in Healthy Male Subjects (an Open-label, Two-period, Fixed-sequence Trial)
Brief Title: Bioavailability of BI 144807 Given Alone and in Combination With Ketoconazole in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1313.7; 2012-003225-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-10-15; First posted 2012-10-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Healthy
MeSH Terms: interventions — Ketoconazole

ARMS (2):
- BI 144807 (Experimental): subjects receive an oral single dose of BI 144807
  Interventions: Drug: BI 144807
- BI 144807 plus Ketoconazole (Experimental): subjects receive bid ketoconazole plus an oral single dose of BI 144807
  Interventions: Drug: Ketoconazole; Drug: BI 144807

INTERVENTIONS:
Drug: Ketoconazole — Ketoconazole 400 mg / day
  Arms: BI 144807 plus Ketoconazole
Drug: BI 144807 — BI144807 oral solution, intermediate dose
  Arms: BI 144807
Drug: BI 144807 — BI144807 oral solution, intermediate dose
  Arms: BI 144807 plus Ketoconazole

SUMMARY:
This trial investigates the influence of oral ketoconazole on the pharmacokinetics and safety of BI 144807.

ELIGIBILITY:
Inclusion criteria:

1. healthy male subjects

Exclusion criteria:

1. any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity | 0 to 48 hours after administration
Maximum measured concentration of the analyte in plasma | 0 to 48 hours after administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point | 0 to 48 hours after administration

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1313.7.1 Boehringer Ingelheim Investigational Site, Biberach, Germany